CLINICAL TRIAL: NCT00773058
Title: Effect of Treatment With Stress-Doses Glucocorticoid on Mortality in Patients With ARDS and Relative Adrenal Insufficiency
Brief Title: Effect of Treatment With Stress-Doses Glucocorticoid in Patients With Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Dr. QIU Hai-bo, Chinese Medical Association
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QHB-YY 2008
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-01

CONDITIONS: Acute Respiratory Distress Syndrome; Adrenal Insufficiency
Keywords: acute respiratory distress syndrome; glucocorticoid; adrenal insufficiency
MeSH Terms: conditions — Respiratory Distress Syndrome; Adrenal Insufficiency | interventions — Hydrocortisone; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- glucocorticoid+RAI (Active Comparator): stress-dose glucocorticoid treatment, compared to placebo group and ACTH test hints RAI
  Interventions: Drug: hydrocortisone
- placebo + RAI (Placebo Comparator): no glucocorticoid But ATCH test hints RAI
  Interventions: Drug: placebo
- glucocorticoid (Active Comparator): stress-dose glucocorticoid treatment, compared to placebo group and ACTH test does not hint RAI
  Interventions: Drug: hydrocortisone
- placebo (Placebo Comparator): no glucocorticoid But ATCH test does not hint RAI
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: hydrocortisone — hydrocortisone 100mg q8h
  Other Names: glucocorticoid; cortical hormone
  Arms: glucocorticoid; glucocorticoid+RAI
Drug: placebo — normal saline 100ml q8h
  Arms: placebo; placebo + RAI

SUMMARY:
The purpose of this study is to see if stress doses of hydrocortisone improve early outcome in patients who are in early stage of ARDS and with relative adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* within the first 3 days of onset of clinically definite ARDS confirmed by AECC criteria in 1994
* 18 to 85 year old

Exclusion Criteria:

* pregnancy or lactation
* tumor or other immunologic disease
* immunosuppressive drug used
* bone marrow or lung transplantation
* primary or secondary disease of adrenal gland
* hormone used within 3 months
* refusing conventional therapy
* be in other clinical tests within 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite ARDS confirmed by AECC criteria in 1994 | within the first 3 days after surgery onset of ARDS